CLINICAL TRIAL: NCT03303976
Title: Safety and Immunogenicity of a Candidate Bioconjugate Vaccine Against Streptococcus Pneumoniae When Administered to Adult and Elderly Healthy Subjects. A Phase I Randomized Study.
Brief Title: Phase I to Test a New Pneumococcal Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pneumo1
Record Dates: First submitted 2017-09-25; First posted 2017-10-06 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Pneumococcal Pneumonia; Pneumonia, Bacterial
Keywords: pneumococcal vaccine; bioconjugate
MeSH Terms: conditions — Pneumonia, Pneumococcal; Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pneumo1-low dose (Experimental): Arm A: intramuscular injection monovalent bioconjugate pneumococcal vaccine
  Interventions: Biological: Bioconjugate pneumococcal vaccine
- Pneumo1-mid dose (Experimental): Arm B: intramuscular injection monovalent bioconjugate pneumococcal vaccine
  Interventions: Biological: Bioconjugate pneumococcal vaccine
- Pneumo1-target dose (Experimental): Arm C: intramuscular injection monovalent bioconjugate pneumococcal vaccine
  Interventions: Biological: Bioconjugate pneumococcal vaccine
- Pneumovax23 (Active Comparator): Arm D: intramuscular injection multivalent plain polysaccharide vaccine
  Interventions: Biological: Multivalent plain polysaccharide vaccine

INTERVENTIONS:
Biological: Bioconjugate pneumococcal vaccine — Bioconjuagte vaccine against bacterial pneumococcal infection
  Arms: Pneumo1-low dose; Pneumo1-mid dose; Pneumo1-target dose
Biological: Multivalent plain polysaccharide vaccine — Multivalent plain polysaccharide vaccine against bacterial pneumococcal infection
  Arms: Pneumovax23

SUMMARY:
To obtain first-in-human data on a new candidate vaccine against Streptococcus pneumoniae in healthy adult and elderly volunteers.

The study aims to assess the safety and immunogenicity of a bioconjugate investigational vaccine compared to the control group (Pneumovax23).

DETAILED DESCRIPTION:
The study aims to assess the safety and immunogenicity of a new bioconjugate investigational vaccine compared to the control group (Pneumovax23) in a randomised, staggered, 2-steps controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 60 and 70 (inclusive) years of age at the time of vaccination.
* Subject who is willing and able to comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Signed informed consent obtained from the subject.

Exclusion Criteria:

* Health condition that, in the opinion of the investigator, may interfere with optimal participation in the study or place the volunteer at increased risk of adverse events (AEs). Study clinicians, in consultation with the principal investigator, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the medical monitor as appropriate. • Clinically significant abnormalities on physical examination.
* Clinically significant abnormalities on laboratory screening.
* Acute or chronic, clinically significant cardiovascular, pulmonary, hepatic or renal abnormality, diseases and/or insufficiency as determined by physical examination or laboratory tests, in particular: unstable current or history of coronary artery disease or cardiac insufficiency, uncontrolled hypertension, clinically significant history of myocardial infarction, atrial fibrillation, uncontrolled or clinically significant type 2 diabetes, current or history of rheumatoid arthritis or temporal arteritis, current acute or chronic active pulmonary diseases.
* Planned administration of a vaccine not foreseen by the study protocol within 4 weeks before and after the vaccination.
* Previous vaccination with any licensed or investigational pneumococcal vaccine or planned administration of a pneumococcal vaccination not foreseen by the study protocol and during the study period, as reported by subject.
* History of radiologically documented pneumonia or invasive pneumococcal disease (IPD) within 3 years previous to study start, as reported by subject.
* Known hypersensitivity to any components of the pneumococcal conjugate vaccine.
* Previous vaccination with any pseudomonas investigational vaccine as reported by the subject.
* Known or suspected impairment of immunological function, documented Human Immunodeficiency Virus (HIV) infection, asplenia, or history of autoimmune disease.
* History of regular use (>2 weeks) in the last 6 months of immunosuppressive drugs including systemic corticosteroids (e.g. corticosteroids ≥0.5 mg/kg BW/day, excluding inhaled and topical steroid).
* Has a coagulation disorder contraindicating intramuscular vaccination..
* Received or receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation or autoimmune disease.
* Received a blood transfusion or previous treatment with blood products, including immunoglobulins within the 3 months preceding the injection, or is scheduled to receive them within 30 days after vaccination.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 3 months preceding the administration of study vaccine, or planned use during the study period.
* BMI (Body Mass Index) <19 or ≥35.
* Positive blood test for HBsAg, hepatitis C virus (HCV), HIV-1/2.
* History of allergy to any vaccine.
* Use of any antibiotic therapy within 1 week preceding injection.
* Subjects with an elective surgical intervention, planned during the study period.
* History of chronic alcohol consumption and/or drug abuse.
* Blood donation of at least 500 mL blood draw within 3 months preceding injection or planned during the study period as reported by subject.
* Pregnancy or intention to become pregnant as reported by subject.
* Female subjects who are not postmenopausal for at least 2 years.
* Man subjects with a female partner in reproductive age refusing to use contraception methods.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | until one month after injection
  Safety and tolerability of the candidate vaccine as determined by occurrence, severity, relationship, of solicited and unsolicited advers events (AEs) and serious adverse events (SAEs) after injection of the candidate vaccine compared to the control group throughout the study until one month after injection.

SECONDARY OUTCOMES:
Clinical laboratory abnormality measure | change from baseline one week after injection and one month after injection
  Safety of the candidate vaccine by measuring changes in haematological and biochemical safety parameters before injection (baseline) and after vaccine administration, in terms of absolute changes and between groups.
Assess immunogenicity of the candidate vaccine | one month and six months after injection
  Evaluation of antigen-specific antibodies levels and functionality at each time point for all groups in terms of change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leidig, MD, Principal Investigator — CRS Mönchengladbach
Locations (1):
- CRS, Mönchengladbach, Germany

IPD SHARING:
Plan to Share IPD: Undecided